CLINICAL TRIAL: NCT05787964
Title: Systems Biology Analysis of Vaccine-induced Immunity to Infectious Diseases in Healthy Participants and Participants With Cancer
Brief Title: Immunity to Infection in Healthy Participants and Participants With Cancer
Acronym: SYS01
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: SYS01
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Influenza; SARS-CoV-2; Hematologic Malignancy; Solid Tumor
MeSH Terms: conditions — Influenza, Human; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be drawn from participants, and different fractions will be isolated and cryopreserved, including peripheral blood mononuclear cells (PBMCs), plasma, serum, and RNA (in PAXgene tubes).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy participants: Healthy adults aged > 18 years
  Interventions: Procedure: Biological sample collection
- Participants with haematological malignancies: Multiple myeloma patients receiving lenalidomide and smoldering multiple myeloma patients under observation.
  Interventions: Procedure: Biological sample collection
- Participants with solid tumours: Stage IV non-small cell lung cancer patients treated with checkpoint inhibitor therapy +/- chemotherapy.
  Interventions: Procedure: Biological sample collection

INTERVENTIONS:
Procedure: Biological sample collection — Whole blood (blood draw/phlebotomy) will be obtained to proceed with immunologic analysis of samples. Collection of biologic samples will occur up to 12 months.

SUMMARY:
Many cancer patients are highly susceptible to infection and respond poorly to vaccination. This observational study will determine molecular and cellular features of immunity to viral pathogens in participants with cancer and compare them to healthy controls. The aim is to identify how antiviral immunity in participants with cancer differs from that in healthy participants to understand why cancer patients are more susceptible to infections. In this context, the investigators will also evaluate immunity to medically indicated severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and seasonal influenza vaccine received by study participants during standard care (vaccines are not part of the study).

DETAILED DESCRIPTION:
Cancer and its treatments are associated with dysregulated immune systems, and cancer patients are highly susceptible to infections (e.g., influenza, SARS-CoV-2). Importantly, cancer patients often respond poorly to vaccination. The molecular and cellular mechanisms underlying immune dysregulation and poor immunity in cancer patients are manifold, variable among individual patients/conditions, and poorly understood. An in-depth understanding of these mechanisms is essential to identifying novel strategies to prevent infectious diseases and developing individualized therapies.

In this observational study, the investigators will collect blood samples from 200 participants with hematological and oncological malignancies and healthy participants and analyze the cellular and humoral immune status in the context of SARS-CoV-2 and influenza infection and vaccination within these samples using systems biological tools. Medically indicated vaccination against SARS-CoV-2 and influenza during study participation is allowed.

This study aims to (1) examine the fundamental innate, cellular, and humoral immune responses to pathogens that form the basis of immunological memory and (2) identify molecular and cellular mechanisms responsible for the reduced immune immunity to viral pathogens in participants with cancer.

ELIGIBILITY:
Inclusion Criteria:

* You are aged 18 years or older.
* You are able to understand and give informed consent.
* Participants with cancer: you are suffering from cancer
* Healthy participants: you are a healthy individual.

Exclusion Criteria:

* You are unable to give informed consent.
* You have been suffering from an acute infection with fever during the last three days.
* You have a Hb level of less than 9 g/dl.
* You have a human immunodeficiency virus (HIV) or hepatitis C virus (HCV) infection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with cancer will be drawn from the local clinics at the University Hospital Tübingen. Healthy participants will be recruited from university and hospital employees not associated with the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Differences in virus-specific antibody levels | 12 months
  Determination of differences in plasma and serum antibody levels between healthy participants and participants with cancer.
Differences in cytokine levels | 12 months
  Determination of differences in plasma and serum cytokine levels between healthy participants and participants with cancer.
Differences in immune cell composition | 12 months
  Determination of quantitative, phenotypical, and functional differences in immune cells from healthy participants and participants with cancer.
Differences in molecular immune cell makeup | 12 months
  Determination of epigenetic, transcriptional, and proteomic makeup of immune cells from healthy participants and participants with cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lengerke, Ph.D., Study Director — University Hospital Tübingen; Florian Wimmers, Ph.D., Study Director — University Hospital Tuebingen
Locations (1):
- University Hopsital Tuebingen, Tübingen, Baden-Wurttemberg, Germany